CLINICAL TRIAL: NCT06723067
Title: More Time More Milk - Wearable, Wireless Breast Pumps to Increase Accessibility of Milk Expression for NICU Mothers
Brief Title: A Randomized Controlled Trial of Impact of Wearable, Wireless Breast Pumps on Frequency and Efficacy of Milk Expression in Mothers of Premature Infants
Acronym: MTMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005474
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Premature Birth
Keywords: premature birth; lactation
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Wearable wireless pump provided in week one (Other): Provision of a wearable, wireless pump in week one with support from a lactation specialist, standard of care in week two.
  Interventions: Device: Wearable wireless breast pump
- Wearable wireless pump provided in week two (Other): Standard of care in week one, provision of a wearable, wireless pump in week two with support from a lactation specialist.
  Interventions: Device: Wearable wireless breast pump

INTERVENTIONS:
Device: Wearable wireless breast pump — As above

SUMMARY:
A randomized controlled trial of impact of wearable, wireless breast pumps on how often and how much milk mothers of premature infants can pump.

DETAILED DESCRIPTION:
Randomized, controlled crossover study design. Non-blinded. Mother of infants born at or below 29+6 weeks of gestation will be eligible once their infant is 28 or more days old. Mothers will be provided with a wearable, wireless breast pump in addition to their usual hospital grade pump. Wireless pumps can be used while cuddling their baby, driving too and from the hospital, caring for other children, etc.

ELIGIBILITY:
Inclusion Criteria:

* Mother of infant born at 29+6 weeks or below
* Mother still pumping at 4 weeks since birth

Exclusion Criteria:

* Current use of mothers own wearable pump

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of pumping sessions per day | 7 days
  Number of milk pumping sessions per day

SECONDARY OUTCOMES:
Volume of milk pumped per day | 7 days
  Volume of breast milk pumped per day
Percentage of required volume pumped | 7 days
  Percentage of infants daily required milk volume which was pumped per day

CONTACTS AND LOCATIONS:
Overall Officials: Alan Groves, Principal Investigator — University of Texas at Austin
Locations (1):
- Ascension Seton Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared at the request of other investigators
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12/02/2024, for 2 years